CLINICAL TRIAL: NCT01111227
Title: Inflammatory Cytokines Profile in Individuals Subjected to Surgical Procedures Using Propofol or Isoflurane.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Upeclin HC FM Botucatu Unesp, São Paulo State University, UNESP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: upeclin/HC/FMB-Unesp-40
Record Dates: First submitted 2010-03-11; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Patients in Good Health
Keywords: cytokines; propofol; isoflurane; flow cytometry; Types of General Anesthesia
MeSH Terms: interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Propofol and isoflurane — Comparison of two anesthetic drugs
  Other Names: Diprivan; isoflurane

SUMMARY:
The aim of this study is to assess the profile of cytokines IL-1beta, IL-6, IL-8, IL-10, IL-12 and TNF-alpha under inhalation anesthesia with isoflurane and intravenous anesthesia with propofol in healthy patients subjected to minimally invasive elective surgeries.

DETAILED DESCRIPTION:
Twenty ASA-I patients, subjected to otorhinolaryngology surgery, were randomly allocated in one group to receive anesthesia with isoflurane 1 MAC (minimum alveolar concentration) (n = 20). Other group with twenty ASA-I patients received propofol 2 to 4 microgram mL-1 (n = 20).

Fentanyl 5 mg kg-1 and rocuronium bromide 0.6 mg kg-1 were also administered to all patients. Venous blood (10 mL) was collected from each patient at each of the following times: before the beginning of surgery and anesthesia (T1), 2 h after the beginning of surgery (T2), and on the day after the anesthetic-surgical procedure (T3).

Plasma concentrations of interleukins IL-1beta, IL-6, IL-8, IL-10 and IL-12 and tumor necrosis factor (TNF-alpha) were measured in each sample through flow cytometry technique by using the method Cytometric Bead Array (CBA). Venous blood samples from fifteen volunteers not subjected to stress were also collected as control, and the same cytokines were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health American Society of Anesthesia status physical I
* Elective minor surgery
* General anesthesia

Exclusion Criteria:

* Smokers
* Alcoholics
* Previous medication or radiation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of cytokines profile | Before surgery and anesthesia, 2h after anesthesia and at the following day of the surgery

SECONDARY OUTCOMES:
Evaluation of pro and anti-inflammatory cytokines | before surgery and anesthesia, 2h after anesthesia and at the following day of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marina Á Mazoti, MsC, Principal Investigator — Department of Pathology, Botucatu Medical School, São Paulo State University, UNESP
Locations (1):
- Botucatu Medical School, UNESP, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Mazoti MA, Braz MG, de Assis Golim M, Braz LG, Dias NH, Salvadori DM, Braz JR, Fecchio D. Comparison of inflammatory cytokine profiles in plasma of patients undergoing otorhinological surgery with propofol or isoflurane anesthesia. Inflamm Res. 2013 Oct;62(10):879-85. doi: 10.1007/s00011-013-0643-y. Epub 2013 Jun 22. PMID 23793449